CLINICAL TRIAL: NCT03186248
Title: Comparison of Short Versus Long Oesophageal Myotomy in Cases With Idiopathic Achalasia: A Randomized Single Blinded Trial
Brief Title: Randomized Clinical Trial Comparing Short Versus Long Oesophageal Myotomy in POEM for Achalasia Cardia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Principal investigator, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AIG- 09/05
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Achalasia Cardia
Keywords: Achalasia cardia; myotomy; Per oral endoscopic myotomy; laparoscopic fundoplication
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Intervention Model Description: Double blind randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Double blind randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short myotomy (Experimental): Per oral endoscopic myotomy extending from 3 cm cephalad to 3 cm distal to EGJ
  Interventions: Procedure: Per oral endoscopic myotomy
- Long myotomy (Active Comparator): Per oral endoscopic myotomy extending from 6-8cm cephalad to and 3 cm distal to EGJ.
  Interventions: Procedure: Per oral endoscopic myotomy

INTERVENTIONS:
Procedure: Per oral endoscopic myotomy — General anesthesia will be administered and an esophagogastroduodenoscopy will be performed. Mucosal incision proximal to the gastroesophageal junction (GEJ) will be identified depending on short or long myotomy. A 1.5- to 2-cm mucosal incision will be performed after raising a submucosal wheal. The endoscope will be inserted to create a submucosal tunnel with a combination of blunt dissection, carbon dioxide insufflation, hydro dissection and careful electrocautery. The tunnel will be extended past the GEJ, 3 cm onto the gastric cardia. after myotomy, the mucosal incision will then be closed using standard endoscopic clips.

SUMMARY:
Aim of this study is to compare the outcomes of a short esophageal myotomy extending from 3 cm cephalad to the EGJ, to 3 cm distal to it with a long esophageal myotomy with an additional proximal extension (at least 6 cm cephalad to the EGJ, to 3 cm distal) for POEM procedures. Principle of POEM is to reduce pressure gradient across LES by Myotomy. Hypothesis is that performing short myotomy will result in similar efficacy in achalasia cardia while reducing the total time taken for the procedure and ultimately will result in less complications.

DETAILED DESCRIPTION:
The primary goal of treatment of achalasia cardia (either LHM or POEM) is to divide the muscle at LES to reduce the pressure so that food bolus can pass down into the esophagus. However, there is little evidence regarding the optimal length of this myotomy for either procedure. During LHM the proximal length of myotomy is extended upto 6-8 cm in esophagus and distally to 3 cm in stomach. There are no data on long term outcomes between differential proximal myotomy lengths. The conventionally the esophageal myotomy is extended to 6-8 cm, this is based on technical considerations, as it is the maximum length that can safely be achieved via a laparoscopic, transhiatal approach. High pressure zone of Esophago gastric junction (EGJ) complex extends for 4 cm on an average with 2 cm on esophageal side. It is hypothesized that If shorter proximal myotomy that ablates just the EGJ complex could achieve the same normalization of EGJ physiology as a longer one, there could be several advantages to this modification. It will take less mediastinal dissection of the esophagus, potentially reducing the chances of esophageal perforation, vagal injury and pleural tears. During POEM, a shorter myotomy would allow for creation of a shorter submucosal tunnel, decreasing operative time along with potentially decreasing the incidence of mucosal perforations, pneumothorax and pneumoperitoneum. Additionally, there is chance that many patients regain some esophageal peristalsis after both LHM and POEM. Patients undergoing POEM for type 1 and type 2 Achalasia cardia will be randomised into 2 groups of short oesophageal (3 cm) and long oesophageal ( 6-8 cm) myotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 and 2 achalasia with eckerd score >3 (0-12 scale achalasia) -.
2. Age 18-75 years.
3. Treatment naïve or history of pneumatic balloon dilatation.
4. Willing and able to comply with the study procedures and provide written informed consent form to participate in the study.

Exclusion Criteria:

1. Type 3 achalasia cardia or any other esophageal motility disorder
2. Previous surgery of the esophagus or stomach
3. Active severe esophagitis
4. Large lower esophageal diverticula
5. Large > 3cm hiatal hernia
6. Sigmoid esophagus
7. Known gastroesophageal malignancy
8. Inability to tolerate sedated upper endoscopy due to cardiopulmonary instability, severe pulmonary disease or other contraindication to endoscopy
9. Cirrhosis with portal hypertension, varices, and/or ascites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Comparison of clinical efficacy between short and long myotomy groups | 1 year
  Clinical success defined as Eckardt score≤3 compared between the two groups

SECONDARY OUTCOMES:
Difference in operating time between short and long esophageal myotomy during POEM | Intra-opeartive
  Operating time defined as time taken from mucosal incision to closure of incision after completion of the procedure. Procedure duration was calculated in both the groups and compared
Intraoperative adverse events | At the time of index procedure
  Adverse events encountered during the procedure will be noted. Clinical success with reference to improvement in eckerd score. Change in LES pressure by Manometry ( Assessed at 1and 3 months) Assessment of Gastro Esophageal Reflux Disease (GERD) by Potential of Hydrogen (pH) -impedance and Endoscopy (Assessed at 1 and 3 months) Change in barium column height on timed barium Esophagogram (Assessed at pre procedure at 1 and 3 months).
LES pressure reduction | 1 and 3 months
  In both the arms reduction in mean LES pressure will be compared at 1 and 3 months
Comparison of changes in Eckardt score | 1, 3 and 12 months
  In both the groups Eckardt score ( based on symptoms of Dysphagia, Chest pain, regurgitation and weight loss) will be compared
Comparison of gastroesophageal Reflux disease (GERD) Rates | 3 months
  Both the groups will under go clinical evaluation, esophagograstroscopy and ph metry
Change in barium column height on barium esophagogram | 1 and 3 months
  In both the groups time barium swallow studies will be done to evaluate the oesophageal emptying at 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: mahiboob sayyed, MD, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Mohan Ramchandani, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No